CLINICAL TRIAL: NCT00860912
Title: Veritas Collagen Matrix Cystocele Repair Study - Postmarketing Protocol #CP1004
Brief Title: Veritas Collagen Matrix Cystocele Repair Study - Postmarketing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: IRB# 85852010
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Pelvic Organ Prolapse
Keywords: Veritas; Cystocele; Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse; Cystocele; Prolapse

STUDY DESIGN:
Intervention Model Description: collagen graft reinforcement
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention: Collagen matrix (Experimental): Cystocele repair: Veritas reinforcing material implanted for reinforcement of cystocele repair with collagen matrix
  Interventions: Procedure: Collagen Matrix
- Native tissue repair (Other): Intervention: Cystocele repair performed: No reinforcing material used and routine performance of a cystocele repair using native tissues.
  Interventions: Procedure: Collagen Matrix

INTERVENTIONS:
Procedure: Collagen Matrix — surgical/reinforcing material
  Other Names: Veritas collagen matrix

SUMMARY:
The purpose of this study is to evaluate the Veritas Collagen Matrix in treating female patients with documented occurence of Pelvic Organ Prolapse as evidenced by a cystocele.

DETAILED DESCRIPTION:
Surgery for cystocele repair to be performed. Native tissue repair to be randomized versus reinforcement with Collagen matrix

.

ELIGIBILITY:
Inclusion Criteria:

* Patient is equal or greater than 18 years old
* Female
* Meets follow-up evaluation time frame
* Understands the nature of the procedure and has provided written informed consent
* Is scheduled to undergo vaginal pelvic reconstructive surgery
* Has > 2nd degree midline cystocele

Exclusion Criteria:

* Presence of severe mucosal ulceration
* Previous pelvic organ prolapse surgery using an implant that will affect the use of the VCM or affect the outcome of the study
* Allergy to bovine material
* Severe mucosal atrophy
* Shortened vaginal length as determined by Investigator
* Pregnant or intends to become pregnant during study
* Has a UTI
* Has vault prolapse < 2nd degree cystocele

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2001-12; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the ability of the VCM to treat pelvic organ prolapse as demonstrated by improvement of cystocele as measured by a comparison of POP-Q scores pre and post surgery | 2 years
  prolapse degree on pelvic exam

SECONDARY OUTCOMES:
To evaluate patient satisfaction as measured by a comparison of Quality of Life questions at baseline and post surgery | 2 years
  subjective satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo W Davila, MD, Principal Investigator — Cleveland Clinic Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guerette NL, Peterson TV, Aguirre OA, VanDrie DM, Biller DH, Davila GW. Anterior repair with or without collagen matrix reinforcement: a randomized controlled trial. Obstet Gynecol. 2009 Jul;114(1):59-65. doi: 10.1097/AOG.0b013e3181a81b41. PMID 19546759